CLINICAL TRIAL: NCT05326438
Title: Cultural Innovations for Recovery in Community-Based Learning Environments (CIRCLE) Phase 3: Testing an Online Learning Community Application
Brief Title: mHealth App for Changing Alcohol Use in Alaska Native American Indian People
Acronym: CIRCLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southcentral Foundation (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-12-056
Record Dates: First submitted 2022-03-15; First posted 2022-04-13 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Alcohol Use Disorder
Keywords: Alaska Native; mHealth app; behavioral interventions; alcohol use disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CIRCLE mHealth app (Experimental): The investigators will trial a modified version of the mHealth app called "Connections" with Alaska Native/American Indian people who want to change the way they use alcohol.
  Interventions: Behavioral: CIRCLE mHealth app

INTERVENTIONS:
Behavioral: CIRCLE mHealth app — For the intervention, participants will be given access to an mHealth sobriety app that has been modified for Alaska Native/American Indian people. The app allows people to track their sobriety, learn new recovery skills, track treatment plans, set reminders, journal about their recovery, and discover helpful videos and testimonials through an extensive resource library that includes culturally meaningful content, graphics, music, videos, recovery tools, and testimonials. Users can also participate in an interactive peer platform and/or participate in group chats to engage participants in facilitated discussions about sobriety, lifestyle changes, cultural content, and Community Reinforcement Approach skill-building.
  Other Names: Connections, created by CHESS Health

SUMMARY:
For many people who have trouble with alcohol, peer support - the opportunity to share challenges, problem-solving strategies, and successes with supportive others - can be helpful. Building on Southcentral Foundation's (SCF's) established learning circles for sobriety support, the goal of this study is to culturally adapt and test the acceptability and feasibility of a smartphone app for sobriety support among Alaska Native and American Indian (AN/AI) people. In Aims 1 and 2 of this study, the investigators used input from patients and providers to culturally adapt a commercially available mHealth app for AN/AI people dealing with alcohol misuse. The investigators then merged culturally relevant content (e.g., stories and music) and skill-building modules based on the Community Reinforcement Approach with the existing informational and peer support features of the Connections app, a product of CHESS Health accessible on smartphones and tablets. The investigators will work with up to 125 SCF patients to assess the acceptability, feasibility, and measurable effects of the culturally-adapted app among AN/AI adults 21 and older, relying on questionnaires and interviews to evaluate the app features and utility.

The study's primary outcome is the feasibility and acceptability of the modified CHESS app for AN/AI people as a tool for sobriety. The secondary outcomes are to examine changes in quality of life, alcohol use and problems, self-efficacy in sobriety, and stages of change over the course of using the app. The investigators will also explore whether alcohol use and problems are mediated by frequency of app use, app satisfaction, and alcohol self-efficacy.

DETAILED DESCRIPTION:
Southcentral Foundation (SCF) has a long history of stakeholder engagement, recognizing that engaged patients seek out information, work collaboratively with providers, and are more likely to demonstrate healthy choices and disease-specific self-management behaviors. SCF has used qualitative methods to identify and meet the changing needs of patients. Building on work in Aim 1 and Aim 2, which provided patient feedback about both the Connections app and the intended measurement tools, work in this Aim will include testing a modified version of the app with SCF patients.

The Connections app supports individuals in recovery by reducing relapse and promoting prosocial engagement. The app allows people to track their sobriety, learn new recovery skills, track treatment plans, set reminders, journal about their recovery, and discover helpful videos and testimonials through an extensive resource library. The app also has a "recovery help button" that can be pressed whenever the participant needs urgent help. Examples of Connections content include motivational talks, meditations, addiction recovery speakers, stress management, and anger management. The study team added additional culturally meaningful content, graphics, music, videos, recovery tools, and testimonials. Connections uses a HIPAA and HITRUST compliant interactive peer platform, which allows users to privately message one another and/or participate in group chats. The investigators will utilize the app's mass messaging and group chat capabilities to engage participants in facilitated discussions that are consistent with the policies, services, and treatment philosophies of SCF. The study team will add additional topics such as sobriety, lifestyle changes, cultural content, and skill-building modules based on the Community Reinforcement Approach.

Participants will be asked to utilize the app for at least 3 months, with a 6-month follow-up. Participation in the study will be entirely voluntary and confidential. The investigators plan to recruit no more than 125 AN/AI adults who report a desire to change their alcohol use patterns. The investigators will attempt to recruit at SCF in such a way as to have adequate representation from urban and rural residing customer-owners. Individuals may or may not be engaged in or have a history of treatment services specifically for alcohol use disorders. The investigators will not access customer-owners' medical records for recruitment purposes. The investigators also plan to interview up to 25 participants at the 6-month mark, gathering qualitative data about their experiences using the app.

Data Analytic Plan:

Interviews will be transcribed verbatim and de-identified prior to analysis. Transcripts will be validated for accuracy and uploaded to ATLAS.ti for data management and coding, with categorical demographic information. Members of the qualitative research team will conduct analysis in four iterative steps: (1) familiarizing themselves with the data, (2) generating or applying a priori and emergent codes to the data, (3) searching for thematic patterns, and (4) searching for demographic patterns. Consistency will be maintained through a shared codebook, team coding of selected transcripts, and regular meetings to discuss and resolve discrepancies.

Data analysis of feasibility and acceptability of the Connections app will include descriptive statistics of counts of interaction with the app and total number of days the app was accessed. Bivariate descriptive statistics will be used to examine differences in feasibility by demographics and baseline observations.

Data analysis for survey data will include descriptive statistics and mixed effects modeling to account for correlation of repeated measures within customer-owner participants for quality of life, alcohol use and problems, self-efficacy in sobriety, and stages of change completed in partnership with our external consultants. As part of this analysis, data will be evaluated for selection bias, and measurement error or misclassification bias that are common challenges in repeated measures and longitudinal public health datasets.

ELIGIBILITY:
Inclusion Criteria (self-reported as):

* Alaska Native/American Indian;
* ≥ 21 years of age;
* Having a desire to change drinking behavior;
* Receiving services at Southcentral Foundation and reside in the Anchorage Service Unit (urban and rural);
* English-speaking;
* Having access to a smartphone or tablet.

Exclusion Criteria (self-reported as):

* Not Alaska Native/American Indian;
* Non-English speaking;
* Having a medical or severe psychiatric condition that the PIs determine would make it difficult for the individual to use the app or participate in the interview;
* Not having access to a smartphone or tablet (e.g., iPad, Kindle Fire, etc.).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of the app | 6 months post app use
  Through qualitative interviews, determine the feasibility and acceptability of the Connections app with Alaska Native and American Indian people to modify drinking behavior. 25 participants will be interviewed after they have trialed the app over a 6 month time period.
Changes in alcohol and drug use over time | Baseline, 3 months after using app, 6 months after using app
  Examine changes in alcohol and drug use with the Alcohol Use Disorders Identification Test - 3 (3 items). The scale is scored from 0-12 (where scores of 0 reflect no alcohol use). The higher the score, the more likely it is that the person's drinking is affecting his/her health and safety; higher scores thus reflect greater use of alcohol and is a worse outcome. All participants will be queried.
Changes in self-efficacy to avoid drinking | Baseline, 3 months after using app, 6 months after using app
  Examine changes in self-efficacy to modify behavior over time of app use using a single item: "How confident are you that you will be able to manage your drinking in the next 90 days, or 3 months?" Scores range from 1 (no confidence) to 10 (very confident). Higher scores indicate greater confidence and better outcome. All participants will be queried.
Changes in alcohol associated problems | Baseline, 3 months after using app, 6 months after using app
  Examine whether problems associated with drinking changes over time using the Short Inventory of Problems - Revised. This questionnaire has 6 items and responses are answered from "0" (never) to "3" (always), with answers ranging from 0 to 18. Lower scores mean fewer problems; higher scores mean greater problems and suggest a worse outcome. All participants will be queried.
Changes in motivation to change alcohol use | Baseline, 3 months after using app, 6 months after using app
  Examine whether readiness for treatment changes over time using the Stages of Change Readiness and Treatment Eagerness Scale (19 items). Lower scores indicate poorer readiness, higher scores indicate better outcome and higher motivation. Scores range from 19 to 95. All participants will be queried.
Changes in quality of life scores | Baseline, 3 months after using app, 6 months after using app
  Examine World Health Organization Quality-of-Life Scale to evaluate physical, psychological, social, environmental changes in quality of life, as well as overall quality of life and health. The 26-item instrument covers four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains quality of life and general health items. Each individual item of the scale is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale. Higher scores indicate better outcome, or better quality of life. All participants will be queried.
Changes in positive and negative affect scores | Baseline, 3 months after using app, 6 months after using app
  Examine positive and negative affect using the short form of the positive and negative affect schedule. There are two subscales, five items for positive affect and five items for negative affect. The scale is answered from "1" for very slightly or not at all to "5" for extreme. Scores on each scale can range from 5 to 25. Lower scores indicate less of this type of affect. Higher positive affect scores is a better outcome for the study; higher negative affect scores is a poorer outcome for the study. All participants will be queried.

CONTACTS AND LOCATIONS:
Overall Officials: Ann D Collier, Ph.D., Principal Investigator — Southcentral Foundation
Locations (1):
- Southcentral Foundation, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bush K, Kivlahan DR, McDonell MB, Fihn SD, Bradley KA. The AUDIT alcohol consumption questions (AUDIT-C): an effective brief screening test for problem drinking. Ambulatory Care Quality Improvement Project (ACQUIP). Alcohol Use Disorders Identification Test. Arch Intern Med. 1998 Sep 14;158(16):1789-95. doi: 10.1001/archinte.158.16.1789. PMID 9738608
- [Result] Hoeppner BB, Kelly JF, Urbanoski KA, Slaymaker V. Comparative utility of a single-item versus multiple-item measure of self-efficacy in predicting relapse among young adults. J Subst Abuse Treat. 2011 Oct;41(3):305-12. doi: 10.1016/j.jsat.2011.04.005. Epub 2011 Jun 22. PMID 21700411
- [Result] Kiluk BD, Dreifuss JA, Weiss RD, Morgenstern J, Carroll KM. The Short Inventory of Problems - revised (SIP-R): psychometric properties within a large, diverse sample of substance use disorder treatment seekers. Psychol Addict Behav. 2013 Mar;27(1):307-14. doi: 10.1037/a0028445. Epub 2012 May 28. PMID 22642856
- [Result] Maisto SA, Conigliaro J, McNeil M, Kraemer K, O'Connor M, Kelley ME. Factor structure of the SOCRATES in a sample of primary care patients. Addict Behav. 1999 Nov-Dec;24(6):879-92. doi: 10.1016/s0306-4603(99)00047-7. PMID 10628520
- [Result] Thompson, E. R. (2007). Development and validation of an internationally reliable short-form of the positive and negative affect schedule (PANAS). Journal of cross-cultural psychology, 38(2), 227-242.
- See also: WHO Quality of Life Scale, BREF version — https://www.who.int/tools/whoqol/whoqol-bref

DOCUMENTS (1):
  • Informed Consent Form (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT05326438/ICF_000.pdf